CLINICAL TRIAL: NCT02528864
Title: Multiparametric Magnetic Resonance Imaging and Metabolomics Approaches to Study Biomarkers for Uterine Malignancy
Brief Title: MRI and Metabolomics Biomarkers for Uterine Malignancy
Acronym: EMCAMRS
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gigin Lin, Department of Radiology, Chang Gung Memorial Hospital
Other Study IDs: 103-7316A3
Record Dates: First submitted 2015-07-29; First posted 2015-08-19 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Uterine Neoplasms
Keywords: biomarker; cancer metabolism; chemical exchange saturation transfer; endometrial cancer; diffusion-weighted imaging; magnetic resonance spectroscopy; uterine malignancy
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Plasma sample preparation for global metabolites analysis and lipidomic analysis:
  2. Urine samples will be diluted with distilled water. Samples are centrifuged at 14,000 g for 5 min, and the supernatants will be collected for LC-MS analysis.
  3. Cellular metabolites extraction: Extraction method will be carried out by the method modified by Munger and Patterson. The medium will be aspirated from culture plates containing cells and 80% methanol (at -80°C) will immediately be added.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal endometrium: Control group (n=30) comprising surgical candidates with normal endometrial tissue will be collected for comparison.
- Endometrial/uterine cancer: 1. 1st year: 50 eligible patients surgical candidates of endometrial cancer with pre-operative imaging and biological samples collected during operation.
  2. 2nd year: Enroll another 50 surgical candidates and complete the data regarding clinical MRS/diffusion-weighted imaging and tissue high resolution MRS. Together with the 50 cancer subjects in the first year there will be in total 100 cancer subjects for analysis.
  3. 3rd year: Collect enough positive events with any myometrial involvement (n=30), cervical stromal invasion (n=10) and nodal metastasis (n=10). Together with the 100 cancer subjects in the first and second years there will be in total 150 cancer subjects for analysis.

SUMMARY:
The aims of this project are: (1) To establish a research platform in order to integrate multiparametric imaging and metabolomics data for uterine malignancy. (2) Identify potential surrogate biomarkers for early diagnosis of endometrial cancer by using multiparametric magnetic resonance imaging and metabolomics approach. (3) To develop surrogate biomarkers for uterine malignancy, in detecting tumor involvement of myometrium, cervix, and lymph nodes. The investigators propose a 3-year research project to prospectively collect data from 150 female patients 20-80 years old, with clinically diagnosed or suspected to have uterine malignancy. An additional control group comprising 30 patients with normal endometrial tissue will be enrolled. Robust magnetic resonance (MR) imaging techniques including MR spectroscopy (MRS), diffusion-weighted imaging and chemical exchange saturation transfer (CEST) imaging will be applied. Biological samples (tissue, blood, urine) will be analyzed by detailed metabolomics approach (high-resolution MRS).

DETAILED DESCRIPTION:
In the 1st year part of this project, the investigators aim to identify the differences between normal endometrium and cancer tissue. Standard conventional MR study plus MRS, diffusion-weighted imaging and CEST sequences will be carried out on 30 eligible surgical candidates for pretreatment clinical assessment.Metabolites in cancer tissue will be collected during operation and analyzed using high resolution MRS, and compared with control group. The primary endpoint of this part is to identify different imaging and metabolomic profiles between normal and cancer subjects. In the 2nd year, the investigators will continue accumulate case number, in order to evaluate the diagnostic accuracy of advanced MR imaging and metabolomics biomarker, in prediction of T staging and myometrial involvement. By the end of 3rd year, the investigators will collect 150 patients, with approximately 20 cases with cervical invasion and 20 cases with nodal metastasis, in order to answer how this approach predicts cervical stromal involvement, nodal and distant metastasis.

The clinical importance of this project is answer the most relevant questions, i.e., prediction of tumor involvement of myometrium, cervix, and lymph nodes. This will be important for understanding the background mechanism of changes identified by MR and 18-F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) /PET, in order to develop novel imaging biomarkers or therapeutic targets. Both molecular imaging and metabolomics are complimentary and share similarities: (1) Comprehensive data representing the information of the living system as a whole (2) information rich data which reflecting the complexity of the biological system (3) ease for longitudinal observation. Metabolomics data provides more details on biochemistry whilst imaging data provides more spatial localization details. A combination of imaging and metabolomics approach would be an ideal tool to develop biomarkers for uterine malignancy. By completion of this project, the investigators expect the most important metabolic biomarkers will be established, and potentially serve as functional tools to guide therapy for patient with uterine malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Female 20 ~ 80 years old.
* Clinically diagnosed or suspected to have uterine malignancy.
* Able to understand and provide signed informed consent.
* Willing to receive standard surgical treatment.

Exclusion Criteria:

* Contraindicated to magnetic resonance study: cardiac pacemaker or cochlear implantation.
* Status post major pelvic surgery, total hip replacement or magnetic substance implantation in the pelvis.
* Significant major systemic disease, such as renal failure, heart failure, stroke, acute myocardial infarction/unstable angina, poor controlled diabetes mellitus, poor controlled hypertension.
* Pregnant or breast-feeding women.
* Moderate to severe dementia.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gigin Lin, MD, PhD, Principal Investigator — Department of Medical Imaging and Intervention, Chang Gung Memorial Hospital
Locations (1):
- Department of Medical Imaging and Intervention, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Y, Wu RC, Lin YC, Huang YL, Lin CY, Lo CJ, Lu HY, Lu KY, Tsai SY, Hsieh CY, Yang LY, Cheng ML, Chao A, Lai CH, Lin G. Endometrial cancer risk stratification using MRI radiomics: corroborating with choline metabolism. Cancer Imaging. 2024 Aug 24;24(1):112. doi: 10.1186/s40644-024-00756-x. PMID 39182135